CLINICAL TRIAL: NCT00990535
Title: Efficacy and Safety of High Dose Regimen of Octreotide LAR in Patients With Neuroendocrine Tumors in Progressive Disease: A Phase II, Open, Multicentric Prospective Study
Brief Title: High Dose Somatostatin Analogues in Neuroendocrine Tumors
Acronym: HIDONET
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Federico II University (Other)
Collaborators: University of Perugia, Faculty of Medicine, Department of Internal Medicine (Other); University of Genova (Other); University Hospital, Udine, Italy (Other)
Responsible Party: Annamaria Colao, Dept of Mol Clin Endocrinol Oncol, University Federico II of Naples
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NeuroendoUnit-6
Record Dates: First submitted 2009-10-05; First posted 2009-10-07 (Estimated); Last update posted 2009-10-07 (Estimated); Status verified 2009-10

CONDITIONS: Respiratory Tract Neoplasms; Thymic Neoplasms; Pancreatic Neoplasms; Gastrointestinal Neoplasms; Multiple Endocrine Neoplasia
Keywords: neuroendocrine tumors; octreotide; somatostatin analogues
MeSH Terms: conditions — Respiratory Tract Neoplasms; Thymus Neoplasms; Pancreatic Neoplasms; Gastrointestinal Neoplasms; Multiple Endocrine Neoplasia; Neuroendocrine Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Octreotide-LAR (Experimental): Patients will receive every 21 days an injection of octreotide-LAR 30 mg until progression is documented.
  Interventions: Drug: Octreotide-LAR

INTERVENTIONS:
Drug: Octreotide-LAR — Octreotide-LAR 30 mg administered every 21 days until progression
  Other Names: Sandostatin-LAR; Longastatina-LAR

SUMMARY:
Octreotide (OCT) is a somatostatin analogue (SSA) available in a long-acting formulation, conventionally administered every 28 days at the maximum dose of 30 mg. Together with lanreotide, it is considered the therapy of choice in the control of endocrine syndromes associated with neuroendocrine tumors (NET)s. A complete or partial clinical response to SSA therapy is generally achieved in at least 50% of the patients with neuroendocrine syndrome. Many studies reported a clinical response in 70-90% of functioning NETs. In about 36-50% of the patients with progressive advanced well differentiated NET (WDNET), a stabilization of disease occurs after treatment with subcutaneous OCT. By developing long-acting slow-release SSA formulation, long-acting OCT (LAR), lanreotide-SR, lanreotide-Autogel, the patient's compliance to SSA therapy was improved and escape from treatment, which was common with the subcutaneous formulation, was avoided. However, rate of objective response was not significantly improved as compared to short-acting SSA. On the other hand, it has to be remarked that long-acting SSA are being used in NET patients at doses correspondent to the low doses of short-acting formulation. The higher commercially available doses of LAR is 30 mg, which is assumed to be comparable to 300 µg of short-acting OCT in the therapy of acromegaly.

Only one study was designed to investigate the use of high-dose LAR (160 mg every 28 days). In this study, objective and hormonal responses in patients with progressive metastatic ileal NET non-responder to standard doses, was significantly elevated. However, this compound has never been commercialized and, of consequence, this first preliminary observation has not been confirmed by further studies.

No systematic studies were performed with the commercially available long-acting SSA used in high-dose treatments. In patients with progressive locally advanced or metastatic NET, increase of the dose or reduction of the interval between injections is a relatively common "empirical" clinical practice, but no studies have been performed to evaluate safety and efficacy of this treatment schedule.

DETAILED DESCRIPTION:
The patient population will include the patients with a histologically documented diagnosis of WDNET, defined according to the last WHO Classification criteria for NET of gastro-entero-pancreatic, bronchial, thymic or other origin; and showing tumor progression under a standard dose treatment with LAR (30 mg every 28 days) for at least 6 months. Progressive disease will be defined as increased tumor size according to RECIST definitions.

ELIGIBILITY:
Inclusion Criteria:

* Well differentiated neuroendocrine tumors in disease progression

Exclusion Criteria:

* Well differentiated neuroendocrine tumors without disease progression
* Patients with intolerance to somatostatin analogues

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2006-01; Primary Completion 2007-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Tumor stabilization | 6 months

SECONDARY OUTCOMES:
Symptoms improvement | 6 months
Decrease of chromogranin-A | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Annamaria Colao, MD, PhD, Principal Investigator — University Federico II of Naples
Locations (1):
- University Federico II of Naples, Naples, Italy